CLINICAL TRIAL: NCT00959192
Title: Phase Iia, Multicenter, Randomized, Third-party Unblinded, Adjuvant-controlled, Multiple Ascending Dose, Safety, Tolerability, And Immunogenicity Trial Of Acc-001 Withqs-21 Adjuvant In Japanese Subjects With Mild To Moderate Alzheimer's Disease.
Brief Title: Safety, Tolerability, And Immunogenicity Study Of ACC-001 In Japanese Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3134K1-2206; B2571009 (Other: Alias Study Number)
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar; saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACC-001 + QS-21 (Experimental): Active vaccine + adjuvant, IM injection, dose of 3, 10 and 30 micrograms, at Day 1, month 1, 3, 6 and 12
  Interventions: Biological: ACC-001; Other: QS-21
- QS-21 (Placebo Comparator): Adjuvant, IM injection, dose 50 micrograms, at Day 1, month 1, 3, 6 and 12
  Interventions: Other: QS-21

INTERVENTIONS:
Biological: ACC-001 — IM injection, dose of 3, 10 and 30 micrograms, at Day 1, month 1, 3, 6 and 12
  Arms: ACC-001 + QS-21
Other: QS-21 — IM injection, dose of 50 micrograms, at Day 1, month 1, 3, 6 and 12
  Arms: ACC-001 + QS-21
Other: QS-21 — IM injection, dose 50 micrograms, at Day 1, month 1, 3, 6 and 12
  Arms: QS-21

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of ACC-001, an investigational vaccine, in subjects with mild to moderate Alzheimer's disease in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Alzheimer's Disease
* Mini-Mental State Examination (MMSE) 16-26

Exclusion Criteria:

* Significant Neurological Disease other than Alzheimer's disease
* Major psychiatric disorder
* Clinically significant systemic illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - Meitetsu Hospital, Aichi
  - Ibaraki Prefectural Central Hospital, Ibaraki
  - Shonan Atsugi Hospital, Kanagawa
  - Kitasato University East Hospital, Kanagawa
  - The Jikei University School of medicine, Tokyo
  - Juntendo University Hospital, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Kanto Ctrl Hp of the Mutual Aid Asso of Public school Teache, Tokyo

REFERENCES:
- [Derived] Arai H, Suzuki H, Yoshiyama T. Vanutide cridificar and the QS-21 adjuvant in Japanese subjects with mild to moderate Alzheimer's disease: results from two phase 2 studies. Curr Alzheimer Res. 2015;12(3):242-54. doi: 10.2174/1567205012666150302154121. PMID 25731629
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3134K1-2206&StudyName=Safety%2C%20Tolerability%2C%20And%20Immunogenicity%20Study%20Of%20ACC-001%20In%20Japanese%20Subjects%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- ACC-001 3 Micrograms + QS-21: A cohort of participants who received intramuscular (IM) injection of active vaccine ACC-001 (3 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
- ACC-001 10 Micrograms + QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (10 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
- ACC-001 30 Micrograms + QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (30 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
- QS-21: A cohort of participants who received IM injection of adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
Period: Overall Study
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Started | 6 | 9 | 9 | 8
Completed | 4 | 8 | 6 | 7
Not Completed | 2 | 1 | 3 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Investigator Request | 1 | 0 | 0 | 0
Not completed — Caregiver Request | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21 | Total
Number analyzed (Participants) | 6 | 9 | 9 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.50 (8.73) | 68.00 (10.34) | 74.33 (6.69) | 64.75 (7.15) | 69.81 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 7 | 25
  Male | 0 | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (AEs) by Severity
Description: Number of participants who experienced mild, moderate, or severe AEs (mild = does not interfere with subject's usual function; moderate = interferes to some extent with subject's usual function; severe = interferes significantly with subject's usual function)
Time Frame: Baseline up to 24 months
Population: The safety analysis population includes all of the randomly assigned participants who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Participants
  Mild | 4 | 7 | 7 | 5
  Moderate | 2 | 1 | 1 | 2
  Severe | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Brain Abnormalities in Magnetic Resonance Imaging (MRI) Data
Description: Number of participants with brain abnormalities in MRI data that are either consistent or not consistent with AD, as determined by radiologists.
Time Frame: Baseline up to 24 months
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- ACC-001 3 Micrograms + QS-21: A cohort of participants who received intramuscular (IM) injection of active vaccine ACC-001 (3 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 3, 6, 9 and 12
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Participants
  Abnormal - inconsistent with AD | 1 | 0 | 2 | 0
  Abnormal - consistent with AD | 6 | 9 | 9 | 8

3. Primary Outcome: Number of Participants With Abnormalities in Neurological Examination
Description: Number of participants with abnormalities in neurological examinations as determined by the investigators. Neurological examinations included Mental Status, Speech, Cranial Nerves (including pupil equality and reactivity), Visual field, Sensory, Motor, Coordination, Gait, Primitive reflexes, Tendon reflexes and Romberg.
Time Frame: Baseline up to 24 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Participants
  Total | 1 | 1 | 0 | 0
  Mental Status | 0 | 0 | 0 | 0
  Speech | 0 | 0 | 0 | 0
  Cranial Nerves | 0 | 0 | 0 | 0
  Visual Field | 0 | 0 | 0 | 0
  Sensory | 1 | 0 | 0 | 0
  Motor | 0 | 0 | 0 | 0
  Coordination | 0 | 0 | 0 | 0
  Gate | 0 | 0 | 0 | 0
  Primitive reflexes | 0 | 0 | 0 | 0
  Tendon reflexes | 0 | 0 | 0 | 0
  Romberg | 0 | 1 | 0 | 0

4. Secondary Outcome: Anti-a-beta IgG Titer at Specified Visits
Description: Geometric mean of anti-a-beta IgG titer from pre-study through Week 104
Time Frame: Baseline up to 24 months
Population: The population for immunogenicity analysis includes all of the randomly assigned participants who took at least one dose of study medication, having the baseline and at least one post baseline immunogenicity evaluation.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Units/mL
  Pre-study (n=6,9,9,8) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 2 (n=6,9,9,8) | 62.2 [35.5 to 109.3] | 65.0 [35.5 to 118.9] | 67.0 [34.1 to 131.8] | 50.0 [50.0 to 50.0]
  Week 4 (n=6,9,9,8) | 107.9 [30.3 to 384.4] | 94.2 [40.1 to 221.1] | 79.0 [27.5 to 227.1] | 50.0 [50.0 to 50.0]
  Week 6 (n=6,9,9,8) | 2106.5 [141.7 to 31312.7] | 4793.2 [1261.0 to 18220.0] | 5702.6 [1181.1 to 17288.0] | 50.0 [50.0 to 50.0]
  Week 8 (n=6,9,9,8) | 1143.3 [108.0 to 12104.3] | 2331.4 [512.2 to 10612.3] | 3423.9 [1182.1 to 9917.0] | 50.0 [50.0 to 50.0]
  Week 10 (n=6,9,9,8) | 979.2 [96.8 to 9903.1] | 1674.9 [369.5 to 7592.9] | 2012.4 [643.4 to 6294.9] | 50.0 [50.0 to 50.0]
  Week 14 (n=6,9,9,8) | 6088.4 [714.5 to 51878.2] | 6286.2 [3923.5 to 10071.6] | 9983.5 [2820.9 to 35333.3] | 50.0 [50.0 to 50.0]
  Week 16 (n=6,9,9,8) | 3860.4 [342.5 to 43507.1] | 4170.4 [2641.8 to 6583.4] | 9228.0 [2930.5 to 29058.2] | 50.0 [50.0 to 50.0]
  Week 24 (n=6,9,9,8) | 1151.5 [165.8 to 7998.4] | 1455.0 [936.2 to 2261.1] | 3903.1 [1151.8 to 13226.8] | 50.0 [50.0 to 50.0]
  Week 28 (n=6,9,7,8) | 8216.5 [1550.5 to 43541.2] | 8929.3 [4466.9 to 17849.8] | 7429.5 [3925.7 to 14060.5] | 50.0 [50.0 to 50.0]
  Week 30 (n=6,9,7,8) | 7218.7 [1438.9 to 36213.5] | 7017.4 [3510.7 to 14026.7] | 6162.2 [3062.2 to 12400.6] | 50.0 [50.0 to 50.0]
  Week 40 (n=5,9,8,8) | 3136.4 [651.2 to 15106.7] | 2706.5 [1358.1 to 5393.9] | 3615.5 [1145.5 to 11411.2] | 50.0 [50.0 to 50.0]
  Week 50 (n=6,8,7,8) | 1854.5 [558.3 to 6159.4] | 1255.8 [656.3 to 2402.9] | 1261.4 [699.2 to 2275.9] | 50.0 [50.0 to 50.0]
  Week 54 (n=5,8,7,7) | 2873.6 [264.8 to 31178.1] | 9636.4 [4558.5 to 20370.7] | 8604.6 [4030.7 to 18368.8] | 50.0 [50.0 to 50.0]
  Week 56 (n=4,8,7,7) | 11006.2 [1617.8 to 74878.3] | 7582.4 [3143.9 to 18286.8] | 6201.5 [2921.4 to 13164.5] | 50.0 [50.0 to 50.0]
  Week 66 (n=4,8,7,7) | 7407.9 [1127.0 to 48693.5] | 3942.5 [1539.4 to 10096.9] | 2452.5 [1442.5 to 4169.7] | 50.0 [50.0 to 50.0]
  Week 78 (n=4,8,6,7) | 5108.6 [1013.9 to 25739.1] | 2465.3 [961.9 to 6318.5] | 1316.3 [645.0 to 2686.1] | 50.0 [50.0 to 50.0]
  Week 91 (n=0,1,1,0) | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 546.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 389.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 104 (n=0,1,1,0) | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 414.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 285.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.

5. Secondary Outcome: Anti-a-beta IgM Titer at Specified Visits
Description: Geotmetric mean of anti-a-beta IgM titer from pre-study through Week 104
Time Frame: Baseline up to 24 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Units/mL
  Pre-study (n=6,9,9,8) | 30.9 [17.9 to 53.6] | 28.2 [21.3 to 37.4] | 25.0 [25.0 to 25.0] | 41.5 [21.8 to 78.8]
  Week 2 (n=6,9,9,8) | 77.1 [17.1 to 347.0] | 92.0 [31.7 to 266.6] | 53.5 [22.5 to 127.6] | 42.4 [21.6 to 83.3]
  Week 4 (n=6,9,9,8) | 108.5 [19.4 to 605.6] | 141.5 [41.6 to 481.5] | 108.5 [41.0 to 286.9] | 43.7 [21.6 to 88.3]
  Week 6 (n=6,9,9,8) | 953.2 [95.7 to 9493.1] | 2988.4 [879.2 to 10157.9] | 2381.4 [662.7 to 8556.9] | 43.0 [21.6 to 85.9]
  Week 8 (n=6,9,9,8) | 848.6 [85.6 to 8414.6] | 2940.1 [812.5 to 10639.6] | 2776.2 [622.2 to 12386.2] | 46.9 [23.7 to 92.9]
  Week 10 (n=6,9,9,8) | 850.8 [147.5 to 4907.8] | 2432.1 [661.4 to 8943.5] | 2323.9 [482.5 to 11192.7] | 36.1 [19.1 to 68.2]
  Week 14 (n=6,9,9,8) | 1487.6 [288.1 to 7682.0] | 2231.0 [728.6 to 6831.2] | 4438.5 [1000.5 to 19689.6] | 37.6 [19.6 to 72.3]
  Week 16 (n=6,9,9,8) | 1503.2 [254.5 to 8880.8] | 2484.8 [797.6 to 7740.9] | 4590.6 [1041.7 to 20230.3] | 40.5 [18.4 to 89.5]
  Week 24 (n=6,9,9,8) | 898.5 [222.1 to 3634.1] | 1421.8 [442.7 to 4565.8] | 2396.4 [643.2 to 8928.8] | 40.1 [18.4 to 87.1]
  Week 28 (n=6,9,7,8) | 885.9 [240.0 to 3270.2] | 3395.8 [1356.5 to 8500.9] | 3592.8 [628.7 to 20531.3] | 42.1 [21.3 to 83.3]
  Week 30 (n=6,9,7,8) | 859.5 [273.2 to 2704.0] | 3729.9 [1286.6 to 10812.9] | 2956.7 [636.6 to 13732.9] | 38.9 [19.4 to 78.2]
  Week 40 (n=5,9,8,8) | 449.0 [110.4 to 1825.7] | 2480.5 [760.2 to 8093.8] | 1967.3 [421.5 to 9183.1] | 37.8 [19.2 to 74.4]
  Week 50 (n=6,8,7,8) | 354.2 [75.6 to 1659.4] | 1330.0 [388.5 to 4553.3] | 1326.8 [233.3 to 7546.2] | 39.9 [17.9 to 88.8]
  Week 54 (n=5,8,7,7) | 680.7 [120.0 to 3861.3] | 2605.4 [862.1 to 7874.2] | 3017.0 [678.8 to 13408.9] | 48.3 [19.2 to 121.1]
  Week 56 (n=4,8,7,7) | 1768.3 [342.4 to 9132.4] | 2570.6 [794.2 to 8320.4] | 3051.9 [618.2 to 15066.0] | 40.5 [16.4 to 100.0]
  Week 66 (n=4,8,7,7) | 1213.0 [244.1 to 6027.2] | 1872.7 [523.3 to 6701.7] | 1825.1 [346.2 to 9621.6] | 46.0 [20.2 to 104.4]
  Week 78 (n=4,8,6,7) | 952.8 [251.0 to 3617.1] | 1650.3 [491.4 to 5542.5] | 844.9 [155.4 to 4594.7] | 48.3 [19.0 to 122.8]
  Week 91 (n=0,1,1,0) | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 219.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 351.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 104 (n=0,1,1,0) | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 154.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 258.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.

6. Other Pre Specified Outcome: The Mean Changes in Alzheimer's Disease Assessment Scale-Cognitive Behavior (ADAS-Cog) Score From Baseline at Week 12, 26, 52, 78 and 104.
Description: The ADAS-Cog is a 12-item,objective measure of cognitive function, consisting of 1) Word Recall, 2) Naming Objects and Fingers, 3) Following Commands, 4) Constructional Praxis, 5) Ideational Praxis, 6) Orientation, 7) Word Recognition, 8) Recall of Test Instructions, 9) Spoken Language Ability, 10) Word-Finding Difficulty, 11) Comprehension of Spoken Language and 12) Concentration/Distractibility. For this study, the ADAS-Cog total score is derived by summing the individual scores from items 1 to 11. Total score ranges from 0 to 70 points, with higher scores indicating a greater degree of impairment.
Time Frame: Baseline up to 24 months
Population: Efficacy analyses were performed on the modified intent-to-treat (mITT) population. The mITT population included all of the randomly assigned participants who took at least one dose of study medication, and had the baseline and at least one post baseline evaluation of the key efficacy variable (ADAS-Cog).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Units on a scale
  Week 12 (n=6,9,9,8) | 0.06 (5.20) | 0.52 (4.39) | 2.93 (4.10) | -0.25 (3.30)
  Week 26 (n=6,9,9,8) | 0.39 (4.38) | -0.41 (5.41) | 3.56 (6.74) | -0.63 (5.76)
  Week 52 (n=5,9,7,8) | 1.87 (8.32) | 0.15 (4.82) | 5.05 (6.68) | 1.04 (7.01)
  Week 78 (n=4,8,6,7) | 0.17 (3.50) | 3.40 (7.08) | 5.39 (3.66) | 2.33 (7.78)
  Week 104 (n=0,1,1,0) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | -4.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 8.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

7. Other Pre Specified Outcome: The Mean Changes in Disability Assessment for Dementia (DAD) Score From Baseline at Week 12, 26, 52,78 and 104.
Description: The DAD is administered through an interview with the caregiver and measures instrumental and basic activities of daily living.
  A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores represent less disability in ADL while lower scores indicate more dysfunction.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 8 | 8
Units on a scale
  Week 12 (n=5,9,7,8) | -4.7 (9.7) | 0.7 (2.6) | 1.5 (5.1) | 1.7 (6.4)
  Week 26 (n=6,9,8,8) | -10.1 (14.5) | -0.2 (11.9) | -4.4 (28.6) | -0.6 (6.5)
  Week 52 (n=5,8,6,8) | -11.2 (20.9) | -3.4 (10.7) | -1.8 (5.1) | -3.1 (9.0)
  Week 78 (n=4,8,5,6) | -0.6 (3.1) | -5.4 (7.7) | 0.5 (6.9) | 3.5 (3.2)
  Week 104 (n=0,1,1,0) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 12.8 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

8. Other Pre Specified Outcome: The Mean Changes in Neuropsychological Test Battery (NTB) Score From Baseline at Week 12, 26, 52 and 78.
Description: The NTB is a composite of nine widely used neuropsychological tests that assess immediate and delayed recall of verbal and visual information, attention, verbal fluency and executive function. The cognitive tests included in the NTB are the Wechsler Memory Scale (WMS) Visual-Paired Associates (immediate and delayed), WMS-Verbal Paired Associates (immediate and delayed), Rey Auditory Verbal Learning Test (immediate and delayed), WMS-Digit Span, Controlled Word Association Test, and Category Fluency Test. The NTB z-score is used for analysis. The z-score for each component is calculated through the following formula: z = (y_visit - y_base)/SD_base, where y_visit is a value at a particular time point and y_base is the average test score, and SD_base is the SD based on all participants' observed baseline scores in the study.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Z-score
  Week 12 (n=6,9,8,8) | 0.023 (0.416) | 0.275 (0.280) | -0.028 (0.282) | 0.227 (0.107)
  Week 26 (n=6,9,9,8) | 0.114 (0.423) | 0.254 (0.353) | -0.081 (0.530) | 0.222 (0.308)
  Week 52 (n=5,9,7,8) | 0.081 (0.288) | 0.211 (0.285) | -0.109 (0.263) | 0.213 (0.416)
  Week 78 (n=4,8,6,7) | -0.088 (0.334) | -0.037 (0.494) | -0.120 (0.442) | 0.246 (0.336)
  Week 104 (n=0,1,1,0) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0.514 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.559 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

9. Other Pre Specified Outcome: The Mean Changes in Mini-Mental State Examination (MMSE) Score From Baseline at Week 4, 8, 12, 16, 26, 30, 40, 52, 78 and 104.
Description: The MMSE is a brief, structured examination of cognitive function. It has a total score of 30 points (0-30), and any score equal to or lower than 26 points indicates cognitive impairment.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Number analyzed (Participants) | 6 | 9 | 9 | 8
Units on a scale
  Week 4 (n=6,9,9,8) | 1.7 (1.5) | 1.3 (1.7) | 1.6 (2.7) | 0.4 (2.3)
  Week 8 (n=6,9,9,8) | 2.2 (3.1) | 0.9 (3.2) | 1.3 (1.7) | 0.9 (2.6)
  Week 12 (n=6,9,9,8) | 0.8 (2.8) | 1.1 (2.7) | 1.1 (2.0) | 1.4 (2.7)
  Week 16 (n=6,9,9,8) | 1.5 (3.4) | 1.3 (2.3) | 2.9 (2.5) | 0.4 (1.8)
  Week 26 (n=6,9,8,8) | 0.3 (3.8) | 0.1 (2.6) | 1.0 (2.8) | -0.1 (1.6)
  Week 30 (n=6,9,8,8) | 0.3 (3.7) | 1.2 (2.4) | 1.6 (2.4) | 0.3 (3.3)
  Week 40 (n=4,9,7,8) | 2.3 (2.2) | 0.8 (3.5) | 0.7 (2.0) | 0.5 (3.2)
  Week 52 (n=5,8,7,7) | 0.4 (4.5) | 1.0 (3.8) | 1.1 (2.1) | 0.6 (2.5)
  Week 78 (n=4,8,6,7) | 1.8 (2.5) | -1.4 (3.9) | -0.3 (1.2) | 0.0 (3.2)
  Week 104 (n=0,1,1,0) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | ACC-001 3 Micrograms + QS-21 | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms + QS-21 | QS-21
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/9 | 9/9 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACC-001 3 Micrograms + QS-21 (N=6) | ACC-001 10 Micrograms + QS-21 (N=9) | ACC-001 30 Micrograms + QS-21 (N=9) | QS-21 (N=8)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Injection site erythema (General disorders) | 2 | 1 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 1 | 2
Injection site swelling (General disorders) | 3 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3 | 3
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Positive Rombergism (Investigations) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.